CLINICAL TRIAL: NCT06362681
Title: Randomized Clinical Trial to Evaluate the Effectiveness of Three Remineralizing Agents on Mineral Density in Permanent Teeth and Molars With Molar Incisor Hypomineralization
Brief Title: Effects of Different Remineralization Agents on Molar Incisor Hypomineralization Defects: a Randomized Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Alvaro García Perez, Dr., Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CF-2023-I-13
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Molar Incisor Hypomineralization
Keywords: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization | interventions — Fluorides; casein phosphopeptide-amorphous calcium phosphate nanocomplex; Fluor Protector

STUDY DESIGN:
Intervention Model Description: The children will be randomly divided into the experiment groups: control (oral hygiene motivation only), fluoride varnish, clinpro white Varnish and pastes containing CPP-ACP and followed up for 24 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: using a block randomization technique in which a computer-generated sequence would be used to assign each participant to a particular group in the allocation ratio of 1:1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group I: control (oral hygiene motivation only), (No Intervention): Participants will be advised to brush their teeth and enamel surfaces three times a day with a 1000 ppm fluoride toothpaste (stabilized Tin Fluoride), for which a 75ml/102g tube will be provided to each participant each time. months to ensure compliance and uniformity.
- Group II: fluoride varnish (Flúor Protector Ivoclar Vivadent) (Experimental): The selected participants will have the fluoride varnish applied once a month for the 24 months of the study. The varnish will only be applied to the teeth and molars with HIM.
  Interventions: Other: Fluoride
- Group III: fluoride varnish (Clinpro White Varnish 3M ESPE) (Experimental): The selected participants will have the fluoride varnish applied once a month for the 24 months of the study. The varnish will only be applied to the teeth and molars with HIM.
  Interventions: Other: Fluoride
- Group IV: CPP-ACP (Experimental): Participants will make a single daily application of 0.3 g of CPP-ACP cream (GC America, MI Paste™ Recaldent®) on the enamel surface. This will be done for 24 months, at night, to maintain prolonged contact of this agent with the surface of the tooth. The night time schedule is chosen because the longer the time in which both CPP-ACP and saliva are kept in the mouth, the more effective the result will be. A measuring spoon will be given to each participant to ensure standardized delivery of 0.3 g of CPP-ACP to each participant's enamel surface.
  Interventions: Other: Fluoride

INTERVENTIONS:
Other: Fluoride — Application of remineralizing agents on teeth and molars with MIH during 24 months of follow-up.
  Other Names: Casein phosphopeptide-amorphous calcium phosphate; Fluor protector; Clinpro White Varnish
  Arms: Group II: fluoride varnish (Flúor Protector Ivoclar Vivadent); Group III: fluoride varnish (Clinpro White Varnish 3M ESPE); Group IV: CPP-ACP

SUMMARY:
The aim of this study was to present a comparative evaluation of the long-term efficacy of fluoride varnish( Flúor protector), Clinpro™ White Varnish and pastes containing CPP-ACP in the remineralization of creamy-white and yellow brown defects in incisors and permanent first molars with Molar Incisor Hypomineralization (MIH) in schoolchildren 6-12 years-old in Mexico.

DETAILED DESCRIPTION:
The study included 208 teeth with yellow-brown or creamy-white defects in children aged 6-12 years who were newly diagnosed with MIH with no substance loss or caries or prior restorative treatment. The children will be randomly divided into the experiment groups: control (oral hygiene motivation only), fluoride varnish, clinpro white Varnish and pastes containing CPP-ACP and followed up for 24 months. The evaluations will be made based on the ICDAS criteria and the measurements which were performed using the laser fluorescence method (DIAGNOdent, KaVo, Biberach, Germany) in the follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Children between 6 to 12 years
* They live in the selected study area
* Have at least one permanent incisor or molar with mild or moderate MIH (creamy white and/or yellow or brown opacities)
* That their parents authorize participation in the study through informed consent.
* No proven or suspected allergy and/or sensitivity to milk protein, as it is a component of the CPP-ACP product.

Exclusion Criteria:

* Defects in enamel development related to syndromes, dental fluorosis, amelogenesis imperfecta, dentinogenesis imperfecta.
* Presence of orthodontic appliances.
* Teeth with MIH with restorations, or severe MIH (affected enamel develops post-eruptive enamel breakdown), or carious lesions classified as score >0 according to the ICDAS.
* Children who do not show cooperation in the use of remineralizing agents.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Mineral Density | 24 months
  evaluate and compare variations in mineral density (MD) using laser induced fluorescence (LF) after applying Fluoride Varnish, Clinpro or Casein phosphopeptide amorphous calcium phosphate on teeth with Molar Incisor Hypomineralization (MIH).

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Garcia Pérez, PhD, Principal Investigator — Universidad Nacional Autonoma de Mexico
Locations (1):
- Alvaro Garcia Pérez, San Pedro Apatlaco, Morelos, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Data supporting the findings of this study will be available upon request to the principal investigator of the study.